CLINICAL TRIAL: NCT00522158
Title: Effects of Achieving Very Low LDL-Cholesterol After Treatment With Statins on Steroidogenesis and Cognition
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Baskent University (Other)
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: KA 05/75
Record Dates: First submitted 2007-08-27; First posted 2007-08-29 (Estimated); Last update posted 2007-08-29 (Estimated); Status verified 2007-08

CONDITIONS: Type 2 Diabetes Mellitus; Cardiovascular Disease; LDL Cholesterol; Cognition
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Cardiovascular Diseases | interventions — Simvastatin; Atorvastatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: simvastatin
Drug: atorvastatin

SUMMARY:
We aimed to compare the effect of achieving an LDL-cholesterol <70 vs an LDL-cholesterol <100 mg/dL with simvastatin or atorvastatin on adrenal and testicular steroidogenesis, and cognition in diabetic patients.

ELIGIBILITY:
Inclusion Criteria:

* patients with controlled type 2 diabetes mellitus with overt CVD
* patients with controlled type 2 diabetes mellitus over the age of 40 years without overt CVD,but with one or more major cardiovascular risk factors

Exclusion Criteria:

* uncontrolled hypertension (systolic blood pressure >180 mm Hg or diastolic blood pressure >95 mm Hg); evidence of active active liver disease or hepatic dysfunction defined as a level of liver transaminases >2 times the upper limit of normal; uncontrolled myocardial ischaemia; congestive heart failure (New York Heart Association classification IIIb or IV); hemodynamically important valvular disease; secondary hypercholesterolemia; gastrointestinal disease that might limit drug absorption or partial ileal bypass; myopathy, or rhabdomyolysis; a known hypersensitivity to statins; using any androgenic, estrogenic, progestogenic, antiandrogenic, or antiestrogenic agents or medications that can alter the gonadal steroid milieu; using systemic immunosuppressants or anticoagulants; plasma creatine kinase levels >50% above the upper limit of normal,transient ischaemic attack or stroke in past,severe hypertriglyceridaemia (fasting triglyceride level ≥350 mg/dl,Currently on psychotropic medications, steroids, opiate analgesics, Known case of major neuropsychiatric illness,Poor cognition at baseline [Mini-Mental State Examination(MMSE) score ≤24],Physically or mentally unable to complete tests, history of other risk factors for hearing loss and/or conventional assessment that presented conductive hearing loss, confirmed by acoustic immittance measurement;presence of non-auditory associated disorders that could lead to long-latency potentials, such as neurological diseases or syndromes

Ages: 40 Years to 85 Years | Sex: All
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Zehra Berberoglu, MD, Principal Investigator — Baskent University Faculty of Medicine